CLINICAL TRIAL: NCT02937558
Title: A Phase 2 Proof-of-Concept Study of CSI-Glucagon™ (Continuous Subcutaneous Glucagon Infusion) to Prevent Hypoglycemia With Lower Intravenous Glucose Infusion Rates in Children up to One Year of Age With Congenital Hyperinsulinism
Brief Title: CSI-Glucagon for Prevention of Hypoglycemia in Children With Congenital Hyperinsulinism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XSGO-CH01; 1R44DK105691-01 (NIH)
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Congenital Hyperinsulinism
Keywords: hypoglycemia
MeSH Terms: conditions — Congenital Hyperinsulinism; Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CSI-Glucagon (Double-Blind Phase - 2 days) (Experimental): Glucagon solution delivered as a continuous subcutaneous infusion via a patch pump at a starting dosage of 5 mcg/kg/hr.
  Interventions: Drug: Glucagon
- Placebo (Double-Blind Phase - 2 days) (Placebo Comparator): Vehicle solution delivered as a 24-hour continuous subcutaneous infusion via a patch pump.
  Interventions: Other: Placebo
- CSI-Glucagon (Open-label Phase - Up to 28 days) (Experimental): Glucagon solution delivered as a continuous subcutaneous infusion via a patch pump at a starting dosage of 5 mcg/kg/hr.
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — Room-temperature-stable, non-aqueous injectable liquid formulation of synthetic glucagon peptide
  Other Names: CSI-Glucagon (continuous subcutaneous glucagon infusion)
  Arms: CSI-Glucagon (Double-Blind Phase - 2 days); CSI-Glucagon (Open-label Phase - Up to 28 days)
Other: Placebo — Isotonic saline
  Arms: Placebo (Double-Blind Phase - 2 days)

SUMMARY:
This is a Phase 2, multi-center, randomized, placebo-controlled, double-blind trial with open-label follow-up designed to assess the efficacy of Xeris Glucagon delivered as a continuous subcutaneous infusion to prevent hypoglycemia with lower intravenous glucose infusion rates in children < 1 year of age with congenital hyperinsulinism.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, placebo-controlled, double-blind (DB) parallel group study with open-label follow-up designed to evaluate the efficacy of CSI-Glucagon™ for the prevention of hypoglycemia with lower IV glucose infusion rates when delivered subcutaneously to patients up to 1 year of age with congenital hyperinsulinism. CSI-Glucagon™ is expected to provide a better inpatient treatment option compared to the current standard of care.

The study will consist of three phases:

1. Baseline Phase: First is a baseline stabilization phase during which concomitant therapy with octreotide and diazoxide will be safely weaned and continuous enteric feed will be held constant to the degree possible, with the only factors varying being meal size and IV glucose infusion rate (GIR) adjusted by a set plasma glucose measurement driven algorithm.
2. Blinded, Randomized Treatment Phase: Following the stabilization phase, subjects will be randomly assigned to blinded treatment with either glucagon or placebo, which will be delivered for up to 48 hours with an OmniPod® infusion pump with the controller set to a starting basal rate for glucagon of 5 μg/kg/hr and GIR adjustments used to maintain euglycemia. After 48 hours of blinded treatment, all subjects will transition to open-label active treatment. However, if GIR reduction from baseline is < 20% at 24 hours, subjects will be transitioned early to the open-label phase.
3. Open-label Treatment Phase: The third study period will involve use of CSI-Glucagon™ to manage blood glucose with minimal GIR for up to 28 days of cumulative exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with hyperinsulinism:

   a. Biochemical; detectable insulin (i.e., ≥1 µIU/L) at time of hypoglycemia (i.e, blood glucose <50 mg/dl), and/or suppressed free fatty acids (FFA), and/or suppressed beta-hydroxybutyrate (BOHB) and/or glycemic response to glucagon at time of hypoglycemia.
2. Absolute necessity of intravenous glucose to prevent hypoglycemia:

   1. Having failed diazoxide therapy as defined by inadequacy of 5 days maximum dose of diazoxide to eliminate the need for IV glucose, not necessarily that diazoxide has no effect.
   2. May be on diazoxide and/or octreotide, but these drugs will be weaned off prior to randomization.
   3. May be on dextrose feeds.
3. Patient may be a participant in other study protocols such as observational studies, as long as no investigational intervention has taken place within 24 hrs. prior to screening.
4. Less than 12 months of age at screening.

Exclusion Criteria:

1. History of allergy to glucagon or excipients in the CSI-Glucagon formulation.
2. Currently receiving, or less than 12 hours removed from IV glucagon treatment that resulted in a best achievable GIR > 8 mg/(kg*min), prior to the start of study drug.
3. Diazoxide naïve or within five days of starting diazoxide.
4. Receiving steroids at doses larger than 20 mg/m2/day (hydrocortisone equivalent).
5. Patients with sepsis.
6. Receiving alpha or beta agonists for blood pressure support.
7. Received an investigational or other study drug within 5 half-lives of drug.
8. Body weight less than or equal to 2.3 kg/5.0 lbs.
9. History of pancreatectomy and GIR < 8 mg/(kg*min) after weaning of all concomitant therapies.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-10; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - UCSF School of Medicine, Division of Pediatric Endocrinology, San Francisco, California
  - Washington University, St. Louis Children's Hospital, St Louis, Missouri
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 5 subjects were randomized to active or placebo treatment during the double-blind phase of the study. All subjects completing double-blind treatment were eligible for open-label in-patient treatment with CSI Glucagon.
Pre-assignment Details: The first enrolled subject was not deemed evaluable for responsive to glucagon based upon prior history of glucagon resistance, per investigator.
Groups:
- CSI-Glucagon: Glucagon solution delivered as a continuous subcutaneous infusion via a patch pump at a starting dosage of 5 mcg/kg/hr.
  Glucagon: Room-temperature-stable, non-aqueous injectable liquid formulation of synthetic glucagon peptide
- Placebo: Vehicle solution delivered as a 24-hour continuous subcutaneous infusion via a patch pump.
  Placebo: Isotonic saline
Period: Double-blind Phase
Arm/Group | CSI-Glucagon | Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Open-label Phase
Arm/Group | CSI-Glucagon | Placebo
Started | 5 | 0
Completed | 5 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSI-Glucagon | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: days] | 25 (12.49) | 78.5 (79.90) | 46.4 (50.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinically Meaningful Reduction in Glucose Infusion Rate (Double-Blind)
Description: Change from baseline in glucose infusion rate (GIR) will be determined for each subject at 24 and 48 hours from the start of blinded treatment. Subjects with a decrease in GIR ≥ 20% at 24 hours, and ≥ 33% at 48 hours will be considered to have had a clinically meaningful treatment response.
Time Frame: Baseline to end of blinded treatment at 24 or 48 hours
Population: Evaluable subjects
Measure: Count of Participants; unit: Participants
Arm/Group | CSI-Glucagon | Placebo
Number analyzed (Participants) | 2 | 2
Participants | 2 | 0

2. Secondary Outcome: Percent Change in GIR (Double-Blind)
Description: The groups will be compared for mean percent change in GIR from baseline to the end of the double-blind study phase.
Time Frame: Baseline to the end of blinded treatment at 24 or 48 hours
Population: Evaluable subjects
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | CSI-Glucagon | Placebo
Number analyzed (Participants) | 2 | 2
% change | -50.1 (4.5) | 1.9 (45.9)

3. Secondary Outcome: Number of Subjects With Clinically Meaningful Reduction in Glucose Infusion Rate (Open-Label)
Description: Change from baseline in glucose infusion rate (GIR) will be determined for each subject at the end of open-label treatment. Subjects with a decrease in GIR ≥ 33% will be considered to have had a clinically meaningful treatment response.
Time Frame: Baseline to the end of open-label treatment at 72 hours
Population: Evaluable subjects
Measure: Count of Participants; unit: Participants
Arm/Group | CSI-Glucagon | Placebo
Number analyzed (Participants) | 4 | 0
Participants | 4 | 0

4. Secondary Outcome: Percent Change in Glucose Infusion Rate (Open-Label)
Description: The groups will be compared for mean percent change in GIR from baseline to the end of the open-label study phase.
Time Frame: Baseline to end of treatment at 72 hours
Population: Evaluable subjects
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | CSI-Glucagon | Placebo
Number analyzed (Participants) | 4 | 0
% change | -51.2 (10.3) |

ADVERSE EVENTS:
Time Frame: From the time of informed consent through last administration of the investigational product, which was a maximum of 72 hours.
Groups:
- CSI-Glucagon (Double-Blind); CSI-Glucagon (Open-Label): Glucagon solution delivered as a continuous subcutaneous infusion via a patch pump at a starting dosage of 5 mcg/kg/hr.
  Glucagon: Room-temperature-stable, non-aqueous injectable liquid formulation of synthetic glucagon peptide
Arm/Group | CSI-Glucagon (Double-Blind) | Placebo | CSI-Glucagon (Open-Label)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT02937558/Prot_SAP_000.pdf